CLINICAL TRIAL: NCT04307264
Title: Development and Validation of CHESS Criteria for the Screening of Varices in Patients With Compensated Advanced Chronic Liver Disease (CHESS2001/APPHA2001)
Brief Title: CHESS Criteria for Varices Screening in Compensated Advanced Chronic Liver Disease (CHESS2001/APPHA2001)
Status: Completed | Type: Observational
Sponsor: Hepatopancreatobiliary Surgery Institute of Gansu Province (Other)
Collaborators: LanZhou University (Other); Tianjin Second People's Hospital (Other); The Sixth People's Hospital of Shenyang (Other); Ankang Central Hospital (Other); Guangxi Zhuang Autonomous Region (Unknown); Dalian Sixth People's Hospital (Unknown); Xingtai People's Hospital (Other); Shanghai Tongji Hospital, Tongji University School of Medicine (Other); Seventh Medical Center of PLA Army General Hospital (Other); Zhujiang Hospital (Other); The Fifth Affiliated Hospital of Zunyi Medical College (Other); Sir Run Run Shaw Hospital (Other); Beijing Tsinghua Changgeng Hospital (Other); The Central Hospital of Lishui City (Other); The Affiliated Third Hospital of Jiangsu University (Unknown)
Responsible Party: Principal Investigator, Xiaolong Qi, Director, Institute of Portal Hypertension, Hepatopancreatobiliary Surgery Institute of Gansu Province
Other Study IDs: CHESS2001
Record Dates: First submitted 2020-03-11; First posted 2020-03-13 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2023-04

CONDITIONS: Compensated Advanced Chronic Liver Disease; Varices Needing Treatment
Keywords: Varices needing treatment; Non-invasive; Liver stiffness; Platelet count

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Overall eligible participants: Eligible participants will receive standard esophagogasrtoduodendoscopy, liver stiffness measurement and serological examination (platelet count, alanine aminotransferase, aspartate aminotransferase, total bilirubin, Prothrombin time, albumin).
  Interventions: Procedure: Esophagogasrtoduodendoscopy, liver stiffness measurement

INTERVENTIONS:
Procedure: Esophagogasrtoduodendoscopy, liver stiffness measurement — Time frame between liver stiffness measurement and esophagogastroduodendoscopy is less than 2 weeks.

SUMMARY:
Variceal hemorrhage is the serious complication in patients with compensated advanced chronic liver disease (cACLD). To evaluate the bleeding risk of varices in cACLD, esophagogastroduodenoscopy (EGD) should be performed. Once identified with medium-large varices, or small varices with red signs or Child-Pugh C class, defined as varices needing treatment (VNT), the patients with cACLD are recommended to receive the non-selective beta blockers or endoscopic variceal ligation per Baveno VI consensus. However, EGD is limited by its invasiveness and uncomfortableness. The Baveno VI criteria, which was validated by 310 patients dominant with hepatitis C virus (55.0%), recommended that EGD could be spared in patients with liver stiffness (LS) < 20kPa and platelet count > 150×10^9 cells/L. Furthermore, the expanded-Baveno VI criteria (LS < 25kPa and platelet count > 110×10^9 cells/L), based on European cohort with hepatitis C virus (62.8%), was able to spare more unnecessary endoscopies than the Baveno VI criteria with VNT missed rate < 5%. Nevertheless, a recent Asian-pacific study indicated that though Baveno VI criteria was able to avoid screening endoscopy with 27.6%, it increased the odds of missing VNT in hepatitis B virus-related cACLD. Notably, this study also suggested that the expanded-Baveno VI criteria was not suited for Asian-pacific cohort with hepatitis B virus as the dominant cause with VNT missed rate > 5%. Our study aims to develop and validate an optimal cutoff value of LS and platelet count (CHESS criteria) to safely avoid more unnecessary endoscopies in patients with hepatitis B virus-dominated cACLD.

DETAILED DESCRIPTION:
Variceal hemorrhage is the serious complication in patients with compensated advanced chronic liver disease (cACLD). To evaluate the bleeding risk of varices in cACLD, esophagogastroduodenoscopy (EGD) should be performed. Once identified with medium-large varices, or small varices with red signs or Child-Pugh C class, defined as varices needing treatment (VNT), the patients with cACLD are recommended to receive the non-selective beta blockers or endoscopic variceal ligation per Baveno VI consensus. However, EGD is limited by its invasiveness and uncomfortableness. The Baveno VI criteria, which was validated by 310 patients dominant with hepatitis C virus (55.0%), recommended that EGD could be spared in patients with liver stiffness (LS) < 20kPa and platelet count > 150×10^9 cells/L. Furthermore, the expanded-Baveno VI criteria (LS < 25kPa and platelet count > 110×10^9 cells/L), based on European cohort with hepatitis C virus (62.8%), was able to spare more unnecessary endoscopies than the Baveno VI criteria (40.0% vs 21.5%, p < 0.001) with VNT missed rate < 5%. Nevertheless, a recent Asian-pacific study indicated that though Baveno VI criteria was able to avoid screening endoscopy with 27.6%, it increased the odds of missing VNT in hepatitis B virus-related cACLD. Notably, this study also suggested that the expanded-Baveno VI criteria was not suited for Asian-pacific cohort with hepatitis B virus as the dominant cause with VNT missed rate > 5%. Our study aims to develop and validate an optimal cutoff value of LS and platelet count (CHESS criteria) to safely avoid more unnecessary endoscopies in patients with hepatitis B virus-dominated cACLD.

ELIGIBILITY:
Inclusion Criteria:

* age 18-75 years;
* confirmed cirrhosis based on liver biopsy or clinical findings;
* without decompensated events (e.g. ascites, bleeding, or overt encephalopathy);
* scheduled to undergo esophagogastroduodenoscopy, and liver stiffness measurement;
* estimated survival time>24 months, and model for end-stage liver disease score<19, and without liver transplant;
* with written informed consent.

Exclusion Criteria:

* contradictions for esophagogastroduodenoscopy;
* accepted primary prevention (non-selective beta blockers or endoscopic variceal ligation);
* Child-Pugh score>9;
* time frame between liver stiffness and esophagogastroduodenoscopy>14 days;
* diagnosed as hepatocellular carcinoma or other hepatobiliary and pancreatic malignancies;
* splenectomy or hepatectomy;
* portal vein thrombosis or cavernous transformation of portal vein;
* pregnancy or unknown pregnancy status.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with compensated advanced chronic liver disease
Sampling Method: Probability Sample
Enrollment: 2000 (Actual)
Dates: Start 2020-03-18 (Actual); Primary Completion 2023-03-17 (Actual); Study Completion 2023-03-17 (Actual)

PRIMARY OUTCOMES:
Accuracy of CHESS criteria | 1 day
  To assess the accuracy of Chinese Portal Hypertension Diagnosis and Monitoring Study Group (CHESS) criteria (optimal cutoff value of liver stiffness and platelet count) to avoid unnecessary endoscopies in patients with compensated advanced chronic liver disease

SECONDARY OUTCOMES:
Accuracy of LSPS model | 1 day
  To assess the accuracy of LSPS model (liver stiffness * spleen diameter to platelet counts) for high-risk varices in patients with compensated advanced chronic liver disease

CONTACTS AND LOCATIONS:
Overall Officials: Jiahong Dong, M.D., Study Chair — Beijing Tsinghua Changgeng Hospital; Xiaolong Qi, M.D., Study Chair — LanZhou University; Liting Zhang, M.D., Principal Investigator — LanZhou University; Lin Zhang, M.D., Principal Investigator — Beijing Tsinghua Changgeng Hospital; Fengmei Wang, M.D., Principal Investigator — Tianjin Second People's Hospital; Ye Gu, M.D., Principal Investigator — The Sixth People's Hospital of Shenyang; Zicheng Jiang, M.D., Principal Investigator — Ankang Central Hospital; Guo Zhang, M.D., Principal Investigator — Guangxi Zhuang Autonomous Region; Yong Zhang, M.D., Principal Investigator — Dalian Sixth People's Hospital; Dengxiang Liu, M.D., Principal Investigator — Xingtai People's Hospital; Li Yang, M.D., Principal Investigator — Shanghai Tongji Hospital, Tongji University School of Medicine; Shuai Wang, M.D., Principal Investigator — Seventh Medical Center of PLA Army General Hospital; Hua Mao, M.D., Principal Investigator — Zhujiang Hospital; Chaohui He, M.D., Principal Investigator — The Fifth Affiliated Hospital of Zunyi Medical College; Weiling Hu, M.D., Principal Investigator — Sir Run Run Shaw Hospital; Shengqiang Zou, M.D., Principal Investigator — The Affiliated Third Hospital of Jiangsu University; Chuxiao Shao, M.D., Principal Investigator — The Central Hospital of Lishui City
Locations (15):
- China (15):
  - Ankang Central Hospital, Ankang
  - Beijing Tsinghua Changgung Hospital, Beijing
  - the Seventh Medical Center of PLA General Hospital, Beijing
  - Dalian Sixth People's Hospital, Dalian
  - Zhujiang Hospital, Guangzhou
  - The First Hospital of Lanzhou University, Lanzhou
  - The Central Hospital of Lishui City, Lishui
  - Guangxi Zhuang Autonomous Region, Nanning
  - Shanghai Tongji Hospital, Shanghai
  - Sixth People's Hospital of Shenyang, Shenyang
  - Tianjin Second People's Hospital, Tianjin
  - Xingtai People's Hospital, Xingtai
  - Sir Run Run Shaw Hospital, Zhejiang
  - The Affiliated Third Hospital of Jiangsu University, Zhenjiang
  - the Fifth Affiliated Hospital of Zunyi Medical University, Zhuhai

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Qi X, Berzigotti A, Cardenas A, Sarin SK. Emerging non-invasive approaches for diagnosis and monitoring of portal hypertension. Lancet Gastroenterol Hepatol. 2018 Oct;3(10):708-719. doi: 10.1016/S2468-1253(18)30232-2. PMID 30215362
- [Background] Wang FS, Fan JG, Zhang Z, Gao B, Wang HY. The global burden of liver disease: the major impact of China. Hepatology. 2014 Dec;60(6):2099-108. doi: 10.1002/hep.27406. Epub 2014 Oct 29. PMID 25164003
- [Background] de Franchis R; Baveno VI Faculty. Expanding consensus in portal hypertension: Report of the Baveno VI Consensus Workshop: Stratifying risk and individualizing care for portal hypertension. J Hepatol. 2015 Sep;63(3):743-52. doi: 10.1016/j.jhep.2015.05.022. Epub 2015 Jun 3. No abstract available. PMID 26047908
- [Background] Maurice JB, Brodkin E, Arnold F, Navaratnam A, Paine H, Khawar S, Dhar A, Patch D, O'Beirne J, Mookerjee R, Pinzani M, Tsochatzis E, Westbrook RH. Validation of the Baveno VI criteria to identify low risk cirrhotic patients not requiring endoscopic surveillance for varices. J Hepatol. 2016 Nov;65(5):899-905. doi: 10.1016/j.jhep.2016.06.021. Epub 2016 Jul 5. PMID 27388923
- [Background] Berzigotti A, Seijo S, Arena U, Abraldes JG, Vizzutti F, Garcia-Pagan JC, Pinzani M, Bosch J. Elastography, spleen size, and platelet count identify portal hypertension in patients with compensated cirrhosis. Gastroenterology. 2013 Jan;144(1):102-111.e1. doi: 10.1053/j.gastro.2012.10.001. Epub 2012 Oct 8. PMID 23058320
- [Background] Ding NS, Nguyen T, Iser DM, Hong T, Flanagan E, Wong A, Luiz L, Tan JY, Fulforth J, Holmes J, Ryan M, Bell SJ, Desmond PV, Roberts SK, Lubel J, Kemp W, Thompson AJ. Liver stiffness plus platelet count can be used to exclude high-risk oesophageal varices. Liver Int. 2016 Feb;36(2):240-5. doi: 10.1111/liv.12916. Epub 2015 Sep 6. PMID 26212020
- [Background] Augustin S, Pons M, Maurice JB, Bureau C, Stefanescu H, Ney M, Blasco H, Procopet B, Tsochatzis E, Westbrook RH, Bosch J, Berzigotti A, Abraldes JG, Genesca J. Expanding the Baveno VI criteria for the screening of varices in patients with compensated advanced chronic liver disease. Hepatology. 2017 Dec;66(6):1980-1988. doi: 10.1002/hep.29363. Epub 2017 Oct 30. PMID 28696510
- [Background] Bae J, Sinn DH, Kang W, Gwak GY, Choi MS, Paik YH, Lee JH, Koh KC, Paik SW. Validation of the Baveno VI and the expanded Baveno VI criteria to identify patients who could avoid screening endoscopy. Liver Int. 2018 Aug;38(8):1442-1448. doi: 10.1111/liv.13732. Epub 2018 Mar 25. PMID 29495113
- [Derived] Huang Y, Li J, Zheng T, Ji D, Wong YJ, You H, Gu Y, Li M, Zhao L, Li S, Geng S, Yang N, Chen G, Wang Y, Kumar M, Jindal A, Qin W, Chen Z, Xin Y, Jiang Z, Chi X, Cheng J, Zhang M, Liu H, Lu M, Li L, Zhang Y, Pu C, Ma D, He Q, Tang S, Wang C, Liu S, Wang J, Liu Y, Liu C, Liu H, Sarin SK, Xiaolong Qi. Development and validation of a machine learning-based model for varices screening in compensated cirrhosis (CHESS2001): an international multicenter study. Gastrointest Endosc. 2023 Mar;97(3):435-444.e2. doi: 10.1016/j.gie.2022.10.018. Epub 2022 Oct 14. PMID 36252870
- [Derived] Huang Y, Zhao L, He R, Li S, Liu C, Qi X, Li J. A strategy for varices screening based on acoustic radiation force impulse combined with platelet (CHESS2001): An alternative of Baveno VI criteria. Hepatol Commun. 2022 Nov;6(11):3154-3162. doi: 10.1002/hep4.2076. Epub 2022 Sep 19. PMID 36121707
- [Derived] Huang Y, Zhang W, Xiang H, Liu Y, Yuan L, Zhang L, Hu S, Xia D, Li J, Gao M, Wang X, Qi X, Peng L, Song Y, Zhou X, Zeng J, Tan X, Deng M, Fang H, Qi S, He S, He Y, Ye B, Wu W, Dang T, Shao J, Wei W, Hu J, Yong X, He C, Bao J, Zhang Y, Zhang G, Ji R, Bo Y, Yan W, Li H, Wang Y, Li M, Wang F, Lian J, Liu C, Cao P, Liu Z, Liu A, Zhao L, Li S, Wu Y, Gu Y, Wang Y, Fang Y, Jiang P, Wu B, Liu C, Qi X. Treatment Strategies in Emergency Endoscopy for Acute Esophageal Variceal Bleeding (CHESS1905): A Nationwide Cohort Study. Front Med (Lausanne). 2022 Apr 27;9:872881. doi: 10.3389/fmed.2022.872881. eCollection 2022. PMID 35572990